CLINICAL TRIAL: NCT04607226
Title: A Translational Approach to Cardiorespiratory-Gated Stimulation of the Auricular Branch of the Vagus Nerve for the Treatment of Major Depression
Brief Title: Effects of Respiratory-Gated Transcutaneous Vagal Nerve Stimulation in Major Depression (Phase 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Ronald Garcia, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2019P003698; 26236 (Other Grant/Funding Number: Brain & Behavior Research Foundation)
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder
Keywords: Transcutaneous Vagus Nerve Stimulation; Cardiac autonomic function; Depressive symptomatology
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Active tVNS - 2 Hz (Experimental): Expiratory-gated transcutaneous vagus nerve stimulation on the left auricle with 2 Hz stimulation frequency
  Interventions: Other: Active transcutaneous vagus nerve stimulation
- Active tVNS - 8 Hz (Experimental): Expiratory-gated transcutaneous vagus nerve stimulation on the left auricle with 8 Hz stimulation frequency
  Interventions: Other: Active transcutaneous vagus nerve stimulation
- Active tVNS - 30 Hz (Experimental): Expiratory-gated transcutaneous vagus nerve stimulation on the left auricle with 30 Hz stimulation frequency
  Interventions: Other: Active transcutaneous vagus nerve stimulation
- Active tVNS - 100 Hz (Experimental): Expiratory-gated transcutaneous vagus nerve stimulation on the left auricle with 100 Hz stimulation frequency
  Interventions: Other: Active transcutaneous vagus nerve stimulation
- Sham tVNS (Sham Comparator): Sham transcutaneous vagus nerve stimulation on the left auricle
  Interventions: Other: Sham transcutaneous vagus nerve stimulation

INTERVENTIONS:
Other: Active transcutaneous vagus nerve stimulation — respiratory-gated non-painful electrical stimulation of the auricle for 30 minutes
  Other Names: Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS); transcutaneous vagus nerve stimulation
  Arms: Active tVNS - 100 Hz; Active tVNS - 2 Hz; Active tVNS - 30 Hz; Active tVNS - 8 Hz
Other: Sham transcutaneous vagus nerve stimulation — stimulation of the auricle for 30 minutes
  Other Names: transcutaneous vagus nerve stimulation
  Arms: Sham tVNS

SUMMARY:
This study will evaluate the short term effects of respiratory-gated transcutaneous vagus nerve stimulation on the regulation of cardiovagal activity, depressive symptomatology and immune function in subjects with major depression and determine the optimal stimulation frequency for this population.

DETAILED DESCRIPTION:
This study will compare the acute effects of respiratory-gated transcutaneous vagus nerve stimulation (tVNS) at different stimulation frequencies and sham stimulation during five sessions within a 2 week period. Heart rate variability (HRV) point process adaptive filtering estimation algorithms will be used to evaluate changes in cardiac autonomic physiology in subjects with major depression in response to tVNS. The effects of tVNS on cardiovagal regulation will be evaluated at rest and in response to an emotion reactivity task. Depression rating scales (Beck's Depression Inventory) will be used to evaluate short term effects of tVNS on depressive symptoms in these subjects. In addition, the study will evaluate the acute effects of the stimulation on serum levels of pro-inflammatory cytokines. The stimulation frequency that produces the greatest regulatory effects on depressive symptoms and physiological variables in this population will be used in a second longitudinal phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent Major Depressive Disorder with a current active depressive episode
* Currently not taking psychiatric medications or on a stable therapeutic dose of psychiatric medication for at least 30 days prior to entering the study

Exclusion Criteria:

* History of cardio-, cerebro-, or peripheral vascular disease, diabetes mellitus, morbid obesity (BMI > 40 kg/m2), kidney or liver failure, history of unexplained fainting spells
* Any psychiatric disorder involving a history of psychosis (e.g. schizophrenia, bipolar disorders, severe personality disorders)
* Any chronic condition affecting movement, speech and/or ability to read or follow written instructions
* Substance use disorder, either mild, moderate, or severe within the past 12 months (excludes nicotine)
* History of suicide attempt within the last year or current active suicidal ideation
* History of a clinically defined neurological disorder including, but not limited to: Any condition likely to be associated with increased intracranial pressure; space occupying brain lesion; History of cerebrovascular accident; Transient ischemic attack within two years; Cerebral aneurysm; Dementia; Parkinson's Disease; Huntington's chorea; or Multiple sclerosis.
* Pregnant or nursing
* Metallic implants or devices contraindicating tVNS

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic function | 1 hour
  Changes in cardiac autonomic function (High Frequency power-Heart Rate Variability) between active and sham tVNS.
Change in depressive symptoms assessed by the Beck Depression Inventory | 1 hour
  Changes from baseline to post-stimulation in the score of the Beck Depression Inventory will be compared between active and sham tVNS. (Beck depression inventory minimum score= 0, maximum score= 63; higher total scores indicate more severe depressive symptoms)

SECONDARY OUTCOMES:
Change in serum levels of pro-inflammatory cytokines | 2 hours
  Changes in serum levels of proinflammatory cytokines (Interleukin 1B, Interleukin 6, Tumor necrosis factor alfa) from baseline to post-stimulation will be assessed and compared between active and sham tVNS

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Garcia, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No